CLINICAL TRIAL: NCT00569699
Title: Phase II Trial of Combination Therapy With Bevacizumab and S-1 in Elderly Patients With Unresectable or Recurrent Colorectal Cancer (BASIC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01023019
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Colorectal Cancer
Keywords: S-1; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — S 1 (combination); Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): S-1, Bevacizumab
  Interventions: Drug: S-1, Bevacizumab

INTERVENTIONS:
Drug: S-1, Bevacizumab — S-1 is administered orally on days 1 to 28 of a 42-day cycle. Patients are assigned on the basis of body surface area (BSA) to receive one of the following oral doses twice daily: 40 mg (BSA <1.25 m2), 50 mg (BSA >1.25 to <1.50 m2), or 60 mg (BSA >1.50 m2).
  Bevacizumab 5 mg/kg (body weight) is administered by intravenous infusion on days 1, and 15.

SUMMARY:
The purpose of this study is to determine whether S-1 and bevacizumab are safe in the treatment of unresectable or recurrent colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal carcinoma with inoperable, locally advanced, or metastatic disease, not amenable to curative therapy
2. Measurable disease or non-measurable but assessable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST)
3. Patients with no previous treatment (radiotherapy or chemotherapy). Patients who have received postoperative adjuvant chemotherapy are eligible if relapse is diagnosed more than 180 days after the end of such treatment.
4. Treatment with FOLFIRI and FOLFOX is not indicated.
5. Age >65 years
6. Life expectancy of at least 3 months
7. ECOG PS of 0, 1, or 2
8. Adequate function of major organs as defined below:

   1. Hemoglobin >9.0 g/dL
   2. White blood cell count >3,500/mm3, <12,000/mm3
   3. Neutrophil count >1,500/mm3
   4. Platelet count >100,000/mm3
   5. Total bilirubin <1.5 mg/dL
   6. AST and ALT <100 U/L (<200 U/L in patients with liver metastasis)
   7. Serum creatinine <1.2 mg/dL
   8. Creatinine clearance estimate by the Cockcroft-Gault method >50 mL/min
9. Able to take capsules orally.
10. No electrocardiographic abnormalities within 28 days before enrollment that would clinically preclude the execution of the study, as judged by the investigator.
11. Voluntary written informed consent.

Exclusion Criteria:

1. Serious drug hypersensitivity or a history of drug allergy
2. Active double cancer
3. Active infections (e.g., patients with pyrexia of 38℃ or higher)
4. Uncontrolled hypertension
5. Serious complications (e.g., pulmonary fibrosis, interstitial pneumonitis, heart failure, renal failure, hepatic failure, or poorly controlled diabetes)
6. Moderate or severe ascites or pleural effusion requiring treatment
7. Watery diarrhea
8. Treatment with flucytosine
9. Metastasis to the CNS
10. Pregnant women, possibly pregnant women, women wishing to become pregnant, and nursing mothers. Men who are currently attempting to conceive children.
11. Severe mental disorder
12. Continuous treatment with steroids
13. Urine dipstick for proteinuria should be <2+
14. Thrombosis, cerebral infarction, myocardial infarction, or pulmonary embolism
15. Major surgical procedure, open biopsy, or clinically significant traumatic injury within 4 weeks
16. Long-term daily treatment with aspirin (>325 mg/day)
17. History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding
18. Judged ineligible for participation in the study by the investigator for safety reasons.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival | every course for first three courses, then every other course

SECONDARY OUTCOMES:
Safety, Response rate, Time to progression, Time to treatment failure, Overall survival, Treatment situation | any time

CONTACTS AND LOCATIONS:
Overall Officials: Hiroya Takiuchi, Principal Investigator — Osaka Medical College Hospital
Locations (1):
- Osaka Medical College Hospital, Takatsuki, Osaka, Japan